CLINICAL TRIAL: NCT06754670
Title: Hypophosphatemia in Wean
Brief Title: Effect of Hypophosphatemia on Neuro-excursion Efficiency During Mechanical Ventilator Weaning
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Shitong Diao, Principal Investigator, Peking Union Medical College
Other Study IDs: K6646
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation; Weaning Failure; Hypophosphatemia
MeSH Terms: conditions — Hypophosphatemia | interventions — alpha-glycerophosphoric acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hypophosphatemia group: On the day of weaning, the patient's peripheral blood phosphorus was low(<0.8mmol/ L).
  Interventions: Drug: Sodium Glycerophosphate 216 MG/ML
- Normal phosphorus group: On the day of weaning, the patient's peripheral blood phosphorus was normal.

INTERVENTIONS:
Drug: Sodium Glycerophosphate 216 MG/ML — Low phosphorus patients receive intravenous phosphate supplementation according to the clinical phosphate supplementation protocol at our center: patients with blood phosphorus < 0.4mmol/L receive 40mmol of glycerol phosphate sodium intravenously via infusion or injection over 4-6 hours; patients with blood phosphorus 0.4-0.8mmol/L receive 30mmol of glycerol phosphate sodium intravenously via infusion or injection; Normal phosphorus patients do not require any special treatment.
  Groups: Hypophosphatemia group

SUMMARY:
Hypophosphatemia is a common phenomenon in the ICU, and several retrospective studies have shown that hypophosphatemia is associated with prolonged mechanical ventilation in ICU patients. However, the specific mechanism and causal relationship are not clear. Previous studies have shown that phosphate infusion improves the contraction of the diaphragm induced by exogenous electrical stimulation, but the effect of hypophosphatemia and phosphate supplementation on the pathophysiology in decannulated patients on mechanical ventilation has not been confirmed. The study group hypothesized that hypophosphatemia affects neural conduction function and muscle contraction by affecting ATP synthesis. Correcting hypophosphatemia may improve respiratory muscle strength and potentially improve diaphragmatic neural conduction, ultimately improving the patient's neuromuscular conversion efficiency and facilitating discharge.

1. The attending physician evaluates the patient's ventilator condition daily and meets the disconnection criteria (spontaneous breathing, RSBI < 105 (min*ml)-1, stable hemodynamics: norepinephrine or epinephrine ≤ 0.1μg/kg/min, PEEP ≤ 8cmH2O, FiO2 ≤ 50%, no increase in ventilator support conditions in the past 24 hours, PS 10cmH2O, MAAS score 2-4, pH ≥ 7.30, discontinuation of all sedative medications). After signing an informed consent form, a diaphragm electromyography (EEG) catheter is placed. (The diaphragm EEG catheter is a gastric tube with diaphragm electromyography monitoring function, with the same placement process and risks as a regular gastric tube. There is a small probability of complications such as nasal mucosal damage.)
2. Start CPAP disconnection: Adjust the ventilator PS 10 → 0 cmH2O, and keep the other conditions unchanged. Collect ventilator parameters, diaphragm electromyography (EAdi) parameters, and diaphragm ultrasound parameters at 0, 1, 3, 5, 10, 20, and 30 minutes after the trial begins, and collect the maximum EAdi and diaphragm ultrasound during quiet state.
3. Simultaneously monitor blood inorganic phosphorus, and divide the patients into two groups: the low phosphorus group (<0.8mmol/L) and the control group (0.8-1.4 mmol/L). Low phosphorus patients receive intravenous phosphate supplementation according to the clinical phosphate supplementation protocol at our center [1-5]: patients with blood phosphorus < 0.4mmol/L receive 40mmol of glycerol phosphate sodium intravenously via infusion or injection over 4-6 hours; patients with blood phosphorus 0.4-0.8mmol/L receive 30mmol of glycerol phosphate sodium intravenously via infusion or injection; Normal phosphorus patients do not require any special treatment.
4. 24h after the first CPAP offline, patients in both groups repeated the CPAP offline process, collected related parameters, and measured blood inorganic phosphorus.

ELIGIBILITY:
Inclusion criteria:

age ≥18 years old; Acute respiratory failure, tracheal intubation patients; Invasive ventilator use time ≥48 hours; Clinically determined remission of primary disease, has switched to auxiliary ventilation mode and plans to go offline in the near future.

Exclusion criteria:

patients with severe neuromuscular disease; Patients with central system diseases; Patients using muscle relaxants for more than 48 hours; Patients who have been or are about to be discontinued from life support; Patients with contraindications for gastric tube insertion after esophagogastric fundus varices, digestive tract perforation, and upper digestive tract surgery; Pregnant patients; Ultrasonic window is poor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanical ventilation patients in the weaning stage
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Neural-excursion efficiency | 0,1,3,5,10,20,30minutes after initiation of the SBT
  Diaphragm excursion/diaphragm potential

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided